CLINICAL TRIAL: NCT02786043
Title: An Open-label, Single Arm, Self-controlled Safety and Pharmacokinetics Study to Evaluate the Effect of Propionyl L-carnitine Hydrochloride on Healthy Chinese Subjects by Diet and Multiple-doses
Brief Title: PK Study to Evaluate the Effect of PLC on Healthy Chinese Subjects by Multiple-doses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-201506-PLC-multidose
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Arterial Diseases
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Propionyl-L-Carnitine Hydrochloride

INTERVENTIONS:
Drug: Propionyl-L-Carnitine Hydrochloride — 1g twice a day on first 4 days and 1g/ day on day 5 during Phase III

SUMMARY:
The main objective is to evaluate the effect of Propionyl-L-Carnitine Hydrochloride on clinical pharmacokinetic characteristics and its effect of clinical pharmacokinetic characteristics and safety on healthy Chinese subjects to provide a basis for market authorization registration

DETAILED DESCRIPTION:
This is a single group subject, open-label, self-controlled, 3 periods, multi-doses administration trial. 12 Healthy Chinese volunteers satisfying inclusion criteria were enrolled with equal number of male and female. Each subject goes through a 7-day Run-in period to eliminate the remaining L-carnitine like substance in the food to ensure the baseline level of endougenous L-Carnitien is stable；In period III, during the first 4 days，all healthy subjects take oral Propionyl-L-Carnitine 1g twice daily; on day 5, all healthy subjects take oral Propionyl-L-Carnitine 1g during fasting.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male and female of same proportion. Healthy individuals.
* Age: 19 to 45. Similar age.
* Weight: All subjects need to weigh ≥50 kg. BMI within 19~24 kg/m2. Similar weight between subjects.；
* Blood pressure: SBP 90-139mmHg，DBP 60-89 mmHg；
* Subjects need to understand and agree before the start of trial and signed the informed consent form.
* Subjects have to be able to communicate with the investigator and comply with the trial protocol.

Exclusion Criteria:

Laboratory investigations:

* Any items of safety evaluation index baseline values considered to be clinically significant abnormal by the investigator before the study;
* Hepatitis B surface antigen positive;
* Hepatitis C antibody positive;
* HIV, Syphilis positive;
* During screening or 1st day of trial before drug administration, any ECG abnormality shown

Drug history:

* Taken any drugs that inhibit or induce hepatic metabolism of drug 1 month prior to the trial;
* Taken any drugs within 2 weeks prior to the trial (including prescription drugs, non-prescription drugs and Chinese herbal drugs);

Past medical history and surgical history:

* Past medical history includes structural heart diseases, heart failure, myocardial infarction, angina pectoris, unexplained arrhythmias, Torsade de pointes, ventricular tachycardia, Long QT syndrome or signs and symptoms of Long QT syndrome with family history (evidenced by genetic testing or relatives died of sudden cardiac death at a young age);
* Thyroid disease history or received thyroid surgery;
* Immune diseases history (e.g. thymus disorder history);
* Received surgery within 6 months prior to the trial;
* Serious gastrointestinal disease history (e.g. clinically significant gallbladder disease, known or suspected jaundice, hepatocellular adenoma, hepatic cavernous hemangioma or other hepatic disease);
* Any gastrointestinal, hepatic or renal diseases that affect drug absorption or metabolism within 6 months prior to the trial (excluded regardless resolved);
* Any serious cerebrovascular, respiratory, metabolic and neurological disease history;
* Hematological disease like clotting disorder;
* Tumor history;
* Hypokalemia, hypocalcemia according to the lower limit of reference range provided by the clinical laboratory;

Lifestyle:

* Frequent alcohol intake within 6 months prior to the trial. Over 14 units of alcohol intake per week (1 unit = 17.7ml ethanol, 1 unit = 357 ml 5% alcohol beer or 44ml 40% liquor or 147 ml 12% alcohol wine);
* Smoke >1 cigarette per day within 3 months prior to the trial;
* Drug abuse history and taken drugs (marijuana, cocaine, opiates, benzodiazepines, amphetamines, barbiturates, methadone, tricyclic antidepressants, etc.) within 1 year prior to the trial;
* Drink excess tea, coffee or caffeine-containing drinks (more than 8 cups) per day 2 days before drug administration to 8 days after drug administration;
* Drink grapefruit juice 2 days before drug administration to 8 days after drug administration;

Others:

* Did not consent to use effective contraceptive methods from enrollment to 3 months after drug administration;
* Hypersensitivity including known allergy to the excipients of the drug (microcrystalline cellulose, lactose, silica powder, sodium carboxymethyl starch, magnesium stearate);
* Participated in any other clinical trials within 3 months prior to the trial or planned to participate in any other clinical trials 1 month after enrollment to the last drug administration visit;
* Blood donation within 3 months prior to the trial or planned to donate blood 1 month after enrollment to the last drug administration visit;
* Any food allergy or special request to diet and cannot comply to unified diet;
* Subjects considered to be excluded by investigator;

For female subjects, any following criteria met, apart from criteria above, should also be excluded:

* Taken oral contraceptive pills within 1 month prior to the trial;
* Long term use of estrogen or progesterone injection or implants within 6 months prior to the trial;
* Fertile female subjects without using contraceptive method 2 weeks prior to the trial;
* Fertile female subjects and spouse not consent to use following contraceptive method, condoms, intra-uterine device, etc. after enrollment to 3 months after drug administration;
* During pregnancy or lactation;
* Urine pregnancy test positive;

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Day 3 and 4, 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24h after drug administration on day 5
  To observe area under curve characteristics of Propionyl-L-Carnitine in single or multiple dose groups

SECONDARY OUTCOMES:
cumulative urine excretion rate | 0h-2h, 2-4h, 4-8h, 8-12h, 12-24h after drug administration
  To compare the cumulative urine excretion rate in multiple dose with that in single dose

CONTACTS AND LOCATIONS:
Overall Officials: Heng-yan Qu, Principal Investigator — National Clinical Trial Institution of Affiliated Hospital of Military Medical Sciences